CLINICAL TRIAL: NCT05563922
Title: Organ Preservation Strategy of Total Neoadjuvant Chemoradiotherapy for Early Low Rectal Carcinoma: A Prospective, Exploratory Trial
Brief Title: Organ Preservation Strategy of Total Neoadjuvant Chemoradiotherapy for Low Rectal Carcinoma
Acronym: OP-TNT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-334R
Record Dates: First submitted 2022-09-04; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Rectal Cancer
Keywords: early low rectal cancer;total neoadjuvant treatment;TEM
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All the patients will receive neoadjuvant chemoradiotherapy ( CapOx + radiotherapy) for 2 cycles, one week after chemoradiotherapy, the first evaluation including MRI, colonoscopy, digital rectal examination and serum CEA will be conducted. Patients without tumor progression will continue 4 cycles of chemotherapy （CapOx） until next imaging and serum assessment. After the second assessment, for patients with tumor regression and suitable for TEM will receive local resection otherwise TME. Following treatment strategy will be made base on the final pathology evaluation after surgery, patients with good pathological response (ypT 0-1 without neural vascular invasion) will enter into the follow-up period, otherwise TME will be operated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant concurrent Chemoradiotherapy plus consolidation chemotherapy followed by TEM (Experimental): All the patients will receive neoadjuvant chemoradiotherapy ( CapOx + radiotherapy) for 2 cycles, one week after chemoradiotherapy, the first evaluation including MRI, colonoscopy, digital rectal examination and serum CEA will be conducted. Patients without tumor progression will continue 4 cycles of chemotherapy （CapOx） until next imaging and serum assessment. After the second assessment, for patients with tumor regression and suitable for TEM will receive local resection otherwise TME. Following treatment strategy will be made base on the final pathology evaluation after surgery, patients with good pathological response (ypT 0-1 without neural vascular invasion) will enter into the follow-up period, otherwise TME will be operated.
  Interventions: Combination Product: Total Neoadjuvant Chemoradiotherapy

INTERVENTIONS:
Combination Product: Total Neoadjuvant Chemoradiotherapy — Radiotherapy：45Gy/25F+Boost 50Gy/25F. A total of 45 Gy, 25 fractions of 1.8 Gy, 5 fractions a week
  CapOx:
  Capecitabine 1000mg / m² po bid (1-14 days, 21 days a cycle) Oxaliplatin 130mg / m2 igtt(Day 1, 21 days a cycle) TEM or endoscopic local resection
  Other Names: Total Neoadjuvant Treatment

SUMMARY:
This study aims to evaluate the efficacy and safety of an organ-sparing strategy after neoadjuvant chemoradiotherapy followed by transanal endoscopic microsurgery （TEM） or endoscopic local resection for early low rectal cancer（cT 1-3N0M0）.Besides, the clinical complete response rate and near-clinical complete response rate, organ preservation rate, local recurrence rate, distant metastasis rate and quality of life （QoL） will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* cT1-3N0M0 assessed by CT, MRI and ultrasound colonoscopy
* Rectal adenocarcinoma confirmed by biopsy pathology and the lower edge of the lesion was within 5cm from the anal edge
* Patients who have a strong desire to preserve the anus and are willing to accept neoadjuvant treatment, meanwhile is suitable for the implementation of organ preservation strategy after discussion within the multidisciplinary team of the hospital
* No previous treatment (including endoscopic resection, transanal local resection, radiotherapy, chemotherapy, etc.) before enrollment
* No contraindications to chemoradiotherapy
* No other colorectal organic diseases
* Voluntarily sign the informed consent

Exclusion Criteria:

* Have received previous treatment (including endoscopic resection, transanal local resection, radiotherapy, chemotherapy, etc.) before enrollment
* Patients with concurrent colorectal organic diseases
* Patients with familial polyposis
* Patients with a previous history of colorectal surgery or pelvic radiotherapy that may affect the outcome of this treatment
* Pregnant or lactating women
* The patient or family members could not understand the conditions and objectives of this study
* With a history of uncontrolled epilepsy, central nervous system diseases, or mental disorders, their clinical severity may hinder the signing of an informed consent form or affect their compliance with oral medication
* It is difficult to achieve complete remission base on existing evidence , such as: maximum diameter of cT2/T3 tumor>4cm; suspicious Lateral lymph nodes (maximum diameter) =5mm; baseline CEA≥100; biopsy pathology contains signet ring cell carcinoma mucinous adenocarcinoma; evaluation team determines whether circumferential constrictive tumor should be included or not when necessary Severe heart disease, such as symptomatic coronary heart disease, New York Cardiology Association (NYHA) grade II or above severe congestive heart failure, or severe arrhythmia requiring pharmacological intervention, or a history of myocardial infarction within the last 12 months
* Organ transplantation requires immunosuppressive therapy
* Serious uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases
* The baseline blood routine and biochemical indexes of the subject do not meet the following criteria: hemoglobin ≥90g / L; absolute neutrophil count (ANC) ≥1.5*10^9 / L; platelet ≥100*10^9 / L; ALT and AST≤ 2.5 times normal upper limit; ALP ≤2.5 times normal upper limit; serum total bilirubin <1.5 times normal upper limit; serum normal creatinine"<1 time upper limit; and serum albumin ≥30g / L

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Organ preservation rate at 3 years | 3 years
  Patients with a good pathological response（ypT 0-1 without neural vascular invasion）after neoadjuvant treatment followed by transanal endoscopic microsurgery（TEM）or endoscopic local resection will be offered an organ preservation strategy

SECONDARY OUTCOMES:
Clinical complete response rate after neoadjuvant chemoradiotherapy | 18 weeks
  Define as complete withdrawal of rectal cancer after neoadjuvant radiotherapy and chemotherapy, and no distant metastasis in imaging examination, and no tumor residue in imaging examination and endoscopic biopsy
3-year local recurrence rate | 3 years
  Occurrence of local recurrence in patients with an organ preservation strategy
3-year distant metastases rate | 3 years
  Occurrence of distant metastases in patients with an organ preservation strategy
3-year Disease-free survival（DFS）rates | 3 years
  Disease free survival defined as the time from enrollment to the first documented disease progression of local recurrence or distance metastasis or death due to any cause
3-year overall survival（OS） rates | 3 years
  OS is defined as the time from enrollment to death due to any cause
Quality of life (EORTC-QLQ-C 30, psychological status) | 20 weeks
  Assess QLQ-C30 in patients with an organ preservation strategy
5-year Disease-free survival（DFS）rates | 5 years
  Disease free survival defined as the time from enrollment to the first documented disease progression of local recurrence or distance metastasis or death due to any cause
5-year overall survival（OS） rates | 5 years
  OS is defined as the time from enrollment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wang, M.D., Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No